CLINICAL TRIAL: NCT00004366
Title: Pilot Study of Vestibular Rehabilitation Training for Panic Disorder With Vestibular Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: University of Pittsburgh (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Purpose: Educational/Counseling/Training
Other Study IDs: 199/11944; UPITTS-11760S-950866; 11760S-950866
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2000-06

CONDITIONS: Vestibular Diseases; Agoraphobia; Panic Disorder
Keywords: agoraphobia; anxiety disorder; disease-related problem/condition; neurologic and psychiatric disorders; panic disorder; rare disease; vestibular diseases
MeSH Terms: conditions — Vestibular Diseases; Agoraphobia; Panic Disorder; Anxiety Disorders; Neurologic Manifestations; Mental Disorders; Rare Diseases | interventions — Physical Therapy Modalities

INTERVENTIONS:
Procedure: Physical therapy

SUMMARY:
OBJECTIVES:

I. Evaluate whether vestibular rehabilitation training is of value in reducing anxiety symptoms in patients with panic disorder with or without agoraphobia who have vestibular dysfunction as identified by clinical vestibular tests.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: During the first 4 weeks of study, patients meet with a clinical nurse specialist once a week for approximately 1 hour. During this time, the nature of the anxiety disorder is explained and exposure to previously feared situations is encouraged.

Only patients who remain symptomatic at a stable level following self-exposure will proceed with rehabilitation training.

Patients meet with a physical therapist once a week for 4 weeks to further evaluate the extent of problems associated with balance. Then, patients undergo weekly 1 hour exercises for 8 weeks with the physical therapist, focusing on sensation, head and eye coordination, movement with eyes opened and closed, and gait.

Concurrently, patients meet with the clinical nurse specialist every 4 weeks during and after physical therapy to evaluate the effects of vestibular treatment on anxiety symptoms.

Training is continued if patient is symptomatic; otherwise, patient is discharged from study.

ELIGIBILITY:
* Diagnosed panic disorder with or without agoraphobia
* Vestibular dysfunction, as defined by abnormalities in the caloric and/or rotational tests
* Continued symptomatology after general instructions of the importance of exposure to feared situations
* Absence of acute symptoms of anxiety or depression assessed to need immediate clinical care

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20
Dates: Start 1995-08; Study Completion 2000-05

CONTACTS AND LOCATIONS:
Overall Officials: Rolf G. Jacob, Study Chair — University of Pittsburgh